CLINICAL TRIAL: NCT04998331
Title: Effectiveness and Safety for Re-treatment With Brentuximab-Vedotin (BV) in Patients With Relapsed/Refractory (R/R) CD30+ Malignancies: a Retrospective Medical Chart Review Study in Spain
Brief Title: A Spanish Medical Record Review of Adults With Relapsed or Refractory CD30+ Malignancies When Re-treated With Brentuximab-vedotin
Acronym: BELIEVE
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: C25023; EUPAS44653 (Other: EUPAS)
Record Dates: First submitted 2021-08-06; First posted 2021-08-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hodgkin Disease; Lymphoma, T-Cell, Cutaneous
Keywords: Drug Therapy
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants With CD30-positive Lymphoma: All participants diagnosed with relapsed/refractory (R/R) cHL, CTCL (mycosis fungoides [MF] and cutaneous anaplastic large cell lymphoma [pcALCL]) and sALCL with CD30 positive, and who have previously achieved a CR or PR with BV treatment and subsequently experienced disease progression/relapse and were administered BV retreatment will be observed retrospectively from their initiation of BV treatment until participant's inclusion date in the study or until treatment discontinuation due to toxicities or any cause. All study data will be collected retrospectively from the medical records.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
Participants in the study are adults with CD30-positive malignancies which include classical Hodgkin lymphoma (cHL), cutaneous T-cell lymphoma (CTCL): mycosis fungoides (MF) or primarily cutaneous anaplastic large cell lymphoma (pcALCL), or systemic anaplastic large cell lymphoma (sALCL).

The main aims of the study are as follows:

* to learn about the response rates of participants with relapsed or refractory CD30+ malignancies when re-treated with BV.
* to check for side effects from re-treatment with BV.

The study will take place in approximately 30 hospitals in Spain.

The study doctors will review each participant's medical record at least 6 months after finishing the last dose of re-treatment with BV. This study is about collecting existing information only; participants will not receive treatment or need to visit a study doctor during this study.

DETAILED DESCRIPTION:
This is an observational, non-interventional, retrospective study in participants with R/R CD30 positive cHL, CTCL (MF and pcALCL) and sALCL who have previously achieved a CR or PR with BV treatment and subsequently experienced disease progression were administered BV retreatment.

This study will assess the effectiveness and safety of BV retreatment in the Spanish population in real-world clinical practice. The study will enroll approximately 35 participants.

The data will be collected and recorded from the medical record of participants and also recorded in electronic case report forms (e-CRFs). All the participants will be assigned to a single observational cohort:

• Participants With CD30-positive Lymphoma

This multi-center trial will be conducted in Spain. The overall duration of the study will be approximately 24 months (12 months for medical chart review and 12 until publication submission).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed cHL, CTCL (MF and pcALCL) or sALCL with CD30 positive.
2. Previously treated with BV containing regimen, with evidence of objective response (determined by having achieved CR or PR), and subsequent disease progression or relapse after discontinuing treatment BV retreatment.
3. Participants with data of disease relapse or progression greater than or equal to (>=) 6 months since the last dose of the first treatment with BV.
4. Participant with data available at the participating site since diagnosis of cHL, CTCL (MF and pcALCL) or sALCL.
5. Having received at least, two doses of BV as retreatment and having follow up information available at the site for a minimum period of six months or until death.

Exclusion Criteria:

There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with R/R cHL, CTCL (MF and pcALCL) and sALCL, who have previously experienced a CR or PR with first BV treatment and subsequently experienced disease progression or relapse were administered BV retreatment will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) as Assessed by Investigator Based on Positron Emission Tomography/Computerized Tomography (PET/CT) Status | Up to 6 months post-index date or death, whatever come first
  ORR is the percentage of participants whose best overall response (graded by favorability in the order of clinical response [CR], partial response [PR], stable disease [SD], progressive disease [PD], and not evaluable [NE]) from initiation of BV retreatment to the discontinuation or end of treatment according to response criteria is either CR or PR. ORR will be assessed by investigator using 5-point scale for visually assessing response on the pre and end-of-treatment PET/CT scans. The 5-point scale ranges from: 1 (No uptake), 2 (Uptake less than or equal to [<=] mediastinum), 3 (Uptake greater than [>] mediastinum but <=liver), 4 (Uptake moderately >liver), and 5 (Uptake markedly higher than liver and/no new lesions). Total score ranges from 0-5. In case of unavailability of PET/CT scans, ORR will be assessed as per Revised Criteria for Response Assessment for Malignant Lymphoma. Index date: eligible participants who start BV as retreatment.
Number of Participants Reporting one or More Adverse Events (AEs) | Up to 12 months

SECONDARY OUTCOMES:
Duration of Response (DOR) Based on PET/CT Status | Up to 6 months post-index date or death, whatever come first
  DOR will be calculated as the time (months) from the first documentation of a confirmed CR or PR (whichever is first recorded) to the date of objective PD or death from any cause, whichever is earliest. DOR will be assessed by investigator using 5-point scale for visually assessing response on the pre and end-of-treatment PET/CT scans. The 5-point scale ranges from: 1 (No uptake), 2 (Uptake <=mediastinum), 3 (Uptake >mediastinum but <=liver), 4 (Uptake moderately >liver), and 5 (Uptake markedly higher than liver and/no new lesions). Total score ranges from 0-5. In case of unavailability of PET/CT scans, DOR will be assessed as per Revised Criteria for Response Assessment for Malignant Lymphoma. Index date: eligible participants who start BV as retreatment.
Overall Survival (OS) | From the index date to the date of death from any cause or end of follow-up (up to 6 months)
  OS will be calculated as time (months) from the index date (date of initiation of BV as retreatment) to the date of death from any cause or end of follow-up. Participants alive at the end of the study period will be censored. Index date: eligible participants who start BV as retreatment.
Percentage of Participants With Complete Response Based on PET/CT Status | At the end of retreatment (up to 6 months post-index date or death, whatever come first)
  Complete response will be assessed by investigator using 5-point scale for visually assessing response on the pre and end-of-treatment PET/CT scans. The 5-point scale ranges from: 1 (No uptake), 2 (Uptake <=mediastinum), 3 (Uptake >mediastinum but <=liver), 4 (Uptake moderately >liver), and 5 (Uptake markedly higher than liver and/no new lesions). Total score ranges from 0-5. In case of unavailability of PET/CT scans, complete response will be assessed as per Revised Criteria for Response Assessment for Malignant Lymphoma. Index date: eligible participants who start BV as retreatment.
Time to Clinical Response (CR or PR) | From the index date to the date of documented CR or PR (up to 6 months)
  Time to clinical response will be calculated from the date of index date (date of initiation of BV as retreatment) to the date of documented CR or PR. Index date: eligible participants who start BV as retreatment.
Time to Best Response | From the index date to first documentation of best response documented (up to 6 months)
  Time to best response will be calculated as the time from the index date (date of initiation of BV as retreatment) to first documentation of best response documented. Tumor response will be based on tumour assessments carried out as per local practice. Index date: eligible participants who start BV as retreatment.
Time to Treatment Failure (TTF) | From the index date to first documentation of objective tumor progression or the day of death due to all causes (up to 6 months)
  TTF will be calculated as the time from the index date (date of initiation of BV as retreatment) to first documentation of objective tumor progression or the day of death due to all causes whichever comes earlier. Tumor response will be based on tumour assessments carried out as per local practice. Index date: eligible participants who start BV as retreatment.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (30):
- Spain (30):
  - Hospital General Vega Baja, San Bartolomé, Alicante
  - Hospital Universitario de Alava, Vitoria-Gasteiz, Araba
  - Ico Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Galdakao, Galdakao, Bizkaia
  - Hospital Universitario Donostia, Donostia / San Sebastian, Gipuzkoa
  - Hospital Universitario Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria, Gran Canarias
  - Hospital Universitario Son Espases, Palma de Mallorca, Mallorca
  - Hospital Clinico Universitario Salamanca, Salamanca, Salamnaca
  - Hospital Nuestra Senora de Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital Del Mar, Barcelona
  - Hospital Vall D'Hebron Universitari, Barcelona
  - Hospital Clinic I Provincial De Barcelona, Barcelona
  - Hospital Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario de Jerez, Cadiz
  - Hospital Universitario De La Princesa, Madrid
  - Hospital Sanitas La Zarzuela, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital. Universitario 12 De Octubre, Madrid
  - Hospital Regional Universitario Malaga, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Complejo Hospitalario Universitario de Pontevedra, Pontevedra
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitari I Politecnic La Fe De Valencia, Valencia
  - Hospital Rio Hortega, Valladolid
  - Hospital De Dia Quironsalud Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/6112d601cd353f0032b9205a